CLINICAL TRIAL: NCT05280561
Title: Stress-, Anxiety-, and Cellphone Use-induced Sleep Deficits and Psychological Conditions During the Pandemic and a Potential Complementary Therapy
Brief Title: Stress-induced Sleep Deficits and a Complementary Therapy
Acronym: Sleep-Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jing Liang, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UP-21-00653
Record Dates: First submitted 2022-02-11; First posted 2022-03-15 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Insomnia Due to Anxiety and Fear

STUDY DESIGN:
Intervention Model Description: 288 subjects were recruited for the study. The sample size was based on a prior power analyses using G-Power 3, for a Mixed Model Repeated Measures Analysis of Variance (MMRMA) design, assuming a statistical power of 0.8, moderate effects of the DHM effects on sleep outcomes, and hypothesis tests conducted at a probability value of .05.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHM group (Experimental): This arm is to evaluate DHM effects on the intervention of stress-induced insomnia during the pandemic. DHM granular preparation contains DHM 200 mg plus same excipients as placebo. The 244 participants were taken DHM granular preparation, which was dissolved in ~100 ml water for oral administration, once daily for 20 days.
  Interventions: Dietary Supplement: DHM
- Control group (Placebo Comparator): The placebo contained excipients including extracts of celery, strawberry, oranges, rose, and beet blended in powder form of 1 g
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DHM — DHM is a positive modulator of GABA. We hypothesize the DHM could reduce stress/anxiety induced insomnia during the pandemic
  Arms: DHM group
Dietary Supplement: Placebo — Excipients including extracts of celery, strawberry, oranges, rose, and beet blended in powder form of 1 g
  Arms: Control group

SUMMARY:
The COVID-19 pandemic and social isolation order induced stress/anxiety as well as cellphone dependence. As a result, sleep disruption and mental distress became major health concerns. Gamma-aminobutyric acid type-A receptor (GABAAR) is one of the key players in modulating sleep. Dihydromyricetin (DHM), an herbal compound, plays a role in GABAAR modulation and mitigating anxiety. The investigators' partner in China obtained 288 participants who completed the online survey to gain insight into how stress/anxiety and time spent on cellphones affected sleep and mood. The participants were then enrolled in a randomized placebo-controlled double-blind study to assess the effects of DHM on sleep and improvement on stress/anxiety and cellphone using time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects were recruited in Chengdu and Beijing (city) in China,
* Able and willing to sign informed consent,
* Between 18 -60 years old at time of consent,
* No alcohol, drug, and smoking,
* Not using sleep medication(s) or other psychiatric medications.

Exclusion Criteria:

* Pregnant or Breastfeeding women,
* Currently taking any medications for sleep,
* Reported naps > 3 times per week
* History of sleep apnea,
* Current alcohol, drug, and smoking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 288 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Effect of DHM on sleep duration | 20 days
  Changes in hours of sleep reported as the difference between self-reported hours of sleep before and after DHM or placebo.
Effect of DHM on stress levels | 20 days
  Changes in stress levels reported as the difference between self-reported stress levels before and after DHM or placebo. Stress levels were scaled from 0 to 10, with 10 being the highest stress level.
Effect of DHM on cellphone time | 20 days
  Changes in hours spent on cellphone reported as the difference between self-reported cellphone usage before and after DHM or placebo.
Effect of DHM on feelings after waking up | 20 days
  Changes in negative feelings after waking up, reported as the difference between the self-reported negative feelings before and after DHM or placebo. In the survey, "feelings after waking up" included negative feelings such as tense, lack of motivation, and irritable/angry. To quantify these feelings, a 'Yes' counted as -1 point, a 'No' counted as 0 points, and a 'Not sure' counted as -0.5 points. The sum of these scores were calculated as the total negative feeling after waking up. Lower score (more negative) indicated worse feelings.

CONTACTS AND LOCATIONS:
Locations (1):
- Furise Group Co, Chengdu, Sichuan, China

REFERENCES:
- [Result] Shen Y, Lindemeyer AK, Gonzalez C, Shao XM, Spigelman I, Olsen RW, Liang J. Dihydromyricetin as a novel anti-alcohol intoxication medication. J Neurosci. 2012 Jan 4;32(1):390-401. doi: 10.1523/JNEUROSCI.4639-11.2012. PMID 22219299
- [Result] Liang J, Lopez-Valdes HE, Martinez-Coria H, Lindemeyer AK, Shen Y, Shao XM, Olsen RW. Dihydromyricetin ameliorates behavioral deficits and reverses neuropathology of transgenic mouse models of Alzheimer's disease. Neurochem Res. 2014 Jun;39(6):1171-81. doi: 10.1007/s11064-014-1304-4. Epub 2014 Apr 13. PMID 24728903
- [Result] Silva J, Shao AS, Shen Y, Davies DL, Olsen RW, Holschneider DP, Shao XM, Liang J. Modulation of Hippocampal GABAergic Neurotransmission and Gephyrin Levels by Dihydromyricetin Improves Anxiety. Front Pharmacol. 2020 Jul 9;11:1008. doi: 10.3389/fphar.2020.01008. eCollection 2020. PMID 32742262